CLINICAL TRIAL: NCT02085733
Title: Pro-calcitonin for Early Detection of Septic Arthritis
Status: Completed | Type: Observational
Sponsor: Children's Hospitals and Clinics of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1311-107
Record Dates: First submitted 2014-02-27; First posted 2014-03-13 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Arthritis, Infectious
Keywords: Arthritis, Septic
MeSH Terms: conditions — Arthritis, Infectious

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Possible Septic Arhtritis Patients

SUMMARY:
Background:

Children presenting with non-traumatic joint pain require different treatment depending on the cause of pain. Septic arthritis, which results from a bacterial infection in the joint, often requires a surgical procedure as well as a long course of antibiotics. In contrast, non-septic arthritis is typically treated by management of symptoms and observation. Current diagnostic standards involve microbiologic examination of fluid taken from the affected joint. This procedure can require the patient to be sedated, and the fluid culture analysis can take up to 72 hours. A single laboratory measure that could be easily obtained and quickly analyzed would aid in faster diagnosis, fewer diagnostic tests and lower cost of the diagnostic work-up for this condition.

Recent research on septic arthritis has identified procalcitonin as a potential septic arthritis diagnostic indicator. Procalcitonin (PCT) is secreted by cells in the thyroid at higher levels when the body is facing infection. Procalcitonin levels rise slowly over the first two hours and peak at 24 hours. Levels rise 100-fold in the peripheral blood stream during this time frame. Several studies have indicated PCT is promising potential diagnostic indicator for septic arthritis. Unfortunately, many of these studies have relatively small sample sizes and very few involve pediatric populations. Additional study of PCT and septic arthritis in children will help evaluate the viability of PCT as a diagnostic indicator.

Research Question:

Can serum procalcitonin assist in clinical differentiation between bacterial (septic) and non-bacterial arthritis?

Methods:

Patients presenting with possible septic arthritis in the emergency department will be recruited for this study. Patients who consent to participate will receive the current standard for care, including IV placement, laboratory tests for Erythrocyte sedimentation rate (ESR),white blood cell count (WBC), and C-reactive protein (CRP), x-rays and consultation with pediatric orthopedics. Patients participating in the study will have a portion of the serum collected for typical diagnostic tests analyzed for PCT. Research assistants will collect data from medical records of participants, including lab and imaging results. Patients who do not undergo surgery will be contacted by phone within 7 days of their ED visit to confirm diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. Are 0 - 16 years of age (inclusive)
2. Have a painful, swollen, monoarticular joint
3. Are suspected of having a septic joint
4. Are able to provide assent and parents provide informed consent

Exclusion Criteria:

1. Have reached anatomical maturity indicated by a closed physis in the joint of interest
2. Have neuromuscular and/or metabolic disease
3. Have a chromosomal disorder affecting chromosome 11 in the region of the CALC-1 gene
4. Have received antibiotics within 7 days of the ED visit
5. Are immune deficient
6. Have had surgery in within the last 7 days

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Emergency department patients.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2014-02; Primary Completion 2016-12 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Septic Arthritis | 7 days post ED visit
  The primary outcome will be the presence or absence of septic joint. We will confirm the presence of a septic joint by the growth of bacteria in the synovial fluid or presumed septic arthritis if any of the following three criteria are present: a) > 50,000 white cells in the synovial fluid, b) positive gram stain or c) positive blood culture in the setting of a swollen joint. For patients who do not undergo operative care, we will determine the presence or absence of septic joint by a templated follow-up telephone survey 7 days after enrollment. Patients who do not undergo an operative procedure will be presumed to have non-bacterial causes of their joint pain. Furthermore, culture negative synovial fluid or Lyme positive arthritis will be classified as non-bacterial causes of joint pain.

CONTACTS AND LOCATIONS:
Overall Officials: Anupam B Kharbanda, MD, MSc, Principal Investigator — Children's Minnesota
Locations (1):
- Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota, United States